CLINICAL TRIAL: NCT07030855
Title: Assessing the Efficacy of Elixirium Thymi Compositum in the Treatment of Acute Bronchitis in Pediatric Patients (EXOTIC): A Double-blind, Randomized, Placebo-controlled, Phase 4 Study
Brief Title: Efficacy of Elixirium Thymi Compositum in the Treatment of Acute Bronchitis in Pediatric Patients
Acronym: EXOTIC
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NNGYK/ETGY/03198-4/2025; 2025-520845-61-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Bronchitis
Keywords: Elixirium thymi compositum; thyme; Bronchitis Severity Score; pediatric; bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elixirium thymi compositum (Experimental): For 6-9 years old patients, 6 ml oral solution three times a day for 5 days. For 9-15 years old patients, 8 ml oral solution three times a day for 5 days. For 15-17 years old patients, 10 ml oral solution three times a day for 5 days.
  Interventions: Combination Product: Elixirium thymi compositum (FoNo VIII.)
- Elixirium thymi compositum placebo (Placebo Comparator): A placebo identical in appearance (color) and taste to the investigational product, without the active ingredient (thyme tincture). For 6-9 years old patients, 6 ml oral solution three times a day for 5 days. For 9-15 years old patients, 8 ml oral solution three times a day for 5 days. For 15-17 years old patients, 10 ml oral solution three times a day for 5 days.
  Interventions: Combination Product: Elixirium thymi compositum (FoNo VIII.) placebo

INTERVENTIONS:
Combination Product: Elixirium thymi compositum (FoNo VIII.) — During the study, the dosage is for children and adolescents as follows: 6 ml three times a day for 6-9 years, 8 ml three times a day for 9-15 years, and 10 ml three times a day for 15-17 years.
  Arms: Elixirium thymi compositum
Combination Product: Elixirium thymi compositum (FoNo VIII.) placebo — During the study, the dosage is for children and adolescents as follows: 6 ml three times a day for 6-9 years, 8 ml three times a day for 9-15 years, and 10 ml three times a day for 15-17 years.
  Arms: Elixirium thymi compositum placebo

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Elixirium thymi compositum (Formulae Normales (FoNo) VIII.) compared to a placebo in children between 6 and 17 years old to treat their acute bronchitis. The main question it aims to answer is: Is Elixirium thymi compositum (FoNo VIII.) safe and effective in the treatment of acute bronchitis compared to placebo?

DETAILED DESCRIPTION:
Acute bronchitis is a common disease caused mainly by viral infections. Although there is a standard symptomatic therapy for it, antibiotics are often prescribed, which contributes to an increase in antibiotic resistance. Elixirium thymi compositum (FoNo VIII.) might be an alternative therapeutic option.

The aim is to establish the role of this product by evaluating its clinical efficacy and safety, meanwhile reducing the misuse of antibiotics in treating this condition.

This is a randomized, controlled, double-blinded, two-arm multicenter phase 4 trial. Eligible patients will be pediatric individuals between 6 and 17 years old diagnosed with acute bronchitis. The trial will enroll at least 56 eligible participants with a Total Bronchitis Severity Score (BSS) ranging from 5 to 12 points. Participants will be assigned randomly in a 1:1 ratio to receive either Elixirium thymi compositum at an age-dependent dosage (18-30 ml daily) for 5 days or a placebo with the same concentration and duration.

The trial's primary endpoint is the assessment of symptom improvement in acute bronchitis, as indicated by changes in the BSS score on Day 7. Secondary endpoints include evaluating use of concomitant medications and dietary supplements, safety and tolerability through reported adverse events, and the necessity of antibiotic usage. These secondary endpoints will provide deeper insights into the differences between the treatment and placebo groups. The primary and secondary endpoints will be monitored throughout a follow-up period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. age 6-17 years,
2. diagnosis of acute bronchitis and the Total Bronchitis Severity Score of the patient is between 5-12 points,
3. informed consent form and patient information leaflet signed by the patient and the parent or legal guardian, and
4. no pregnancy, no planned pregnancy, and no breastfeeding.

Exclusion Criteria:

1. allergy to the active ingredients or any other components of Elixirium thymi compositum,
2. hypersensitivity to plants of the Lamiaceae family,
3. chronic respiratory diseases such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease,
4. pneumonia in the last year,
5. a history of recurrent or severe laryngotracheal stenosis due to inflammation,.
6. active or chronic inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis) or infectious enterocolitis,
7. heart failure (New York Heart Association Class II-IV),
8. smoking (the patient currently smokes or has smoked at least one cigarette, cigar, or pipe daily),
9. a diagnosis or history of lung cancer,
10. a history of lung or chest surgery,
11. epilepsy,
12. any viral infection in the last 6-8 weeks,
13. immunostimulant medications, antibiotics, or systemic steroid treatments in the past month,
14. antihistamines, expectorants, or local steroids applied in the last two weeks,
15. hereditary fructose intolerance, glucose-galactose malabsorption, or sucrase-isomaltase deficiency,
16. taking or planning to take hormonal contraceptives within the next 2 weeks
17. chronic liver disease (e.g., cirrhosis) or acute hepatitis.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Bronchitis Severity Score | From enrollment to the end of study at 7 days, measured on Day 0, Day 3 and Day 7.
  The Bronchitis Severity Scale (BSS) is a tool that assesses the five most important symptoms of acute bronchitis: cough, sputum production, wheezing, chest pain on coughing, and dyspnea. The assessment is based on the examiner's clinical judgment and patient feedback. The examiner rates each parameter of the BSS on a 5-point verbal scale from 0 to 4 (0: absent; 1: mild; 2: moderate; 3: severe; 4: very severe). The total BSS score is the sum of the ratings of the five symptoms, with a maximum score of 20.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From enrollment to the end of study at 7 days.
  Any adverse events and concomitant medications during the 7-day period.
Quality of life in acute bronchitis | From enrollment to the end of study at 7 days.
  Quality of life in patients with acute bronchitis was assessed using the Quality of Life Questionnaire, which measures the physical, psychological, and social impact of symptoms during illness. Each question is scored from 1 (absent symptom) to 5 (very severe symptom). Domain scores are calculated as the average of item scores within each domain (Physical: 6 items, Psychological: 7 items, Social: 5 items), resulting in a range of 1 to 5 per domain. The total score, obtained by summing the three domain scores, ranges from 3 (best possible quality of life) to 15 (worst possible quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Noé Medical Center, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available for this study. The informed consent form, in compliance with the EU General Data Protection Regulation (GDPR) and relevant Hungarian laws, specifically informs participants that their data will be handled confidentially, stored anonymously, and presented only in aggregate, anonymized form in any resulting publications. The consent does not include permission for broader sharing of individual-level data outside the study team or approved data processors.

REFERENCES:
- [Background] Saust LT, Bjerrum L, Siersma V, Arpi M, Hansen MP. Quality assessment in general practice: diagnosis and antibiotic treatment of acute respiratory tract infections. Scand J Prim Health Care. 2018 Dec;36(4):372-379. doi: 10.1080/02813432.2018.1523996. Epub 2018 Oct 8. PMID 30296885
- [Background] Braman SS. Chronic cough due to acute bronchitis: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):95S-103S. doi: 10.1378/chest.129.1_suppl.95S. PMID 16428698
- [Background] Cutrera R, Baraldi E, Indinnimeo L, Miraglia Del Giudice M, Piacentini G, Scaglione F, Ullmann N, Moschino L, Galdo F, Duse M. Management of acute respiratory diseases in the pediatric population: the role of oral corticosteroids. Ital J Pediatr. 2017 Mar 23;43(1):31. doi: 10.1186/s13052-017-0348-x. PMID 28335827
- [Background] Gonzales R, Sande MA. Uncomplicated acute bronchitis. Ann Intern Med. 2000 Dec 19;133(12):981-91. doi: 10.7326/0003-4819-133-12-200012190-00014. PMID 11119400
- [Background] Snyder RL, King LM, Hersh AL, Fleming-Dutra KE. Unnecessary antibiotic prescribing in pediatric ambulatory care visits for bronchitis and bronchiolitis in the United States, 2006-2015. Infect Control Hosp Epidemiol. 2021 May;42(5):612-615. doi: 10.1017/ice.2020.1231. Epub 2020 Oct 16. PMID 33059780
- [Background] Wenzel RP, Fowler AA 3rd. Clinical practice. Acute bronchitis. N Engl J Med. 2006 Nov 16;355(20):2125-30. doi: 10.1056/NEJMcp061493. No abstract available. PMID 17108344
- [Background] Gonzales R, Bartlett JG, Besser RE, Cooper RJ, Hickner JM, Hoffman JR, Sande MA; Centers for Disease Control and Prevention. Principles of appropriate antibiotic use for treatment of uncomplicated acute bronchitis: background. Ann Emerg Med. 2001 Jun;37(6):720-7. doi: 10.1067/S0196-0644(01)70091-1. PMID 11385346
- [Background] Kowalczyk A, Przychodna M, Sopata S, Bodalska A, Fecka I. Thymol and Thyme Essential Oil-New Insights into Selected Therapeutic Applications. Molecules. 2020 Sep 9;25(18):4125. doi: 10.3390/molecules25184125. PMID 32917001
- [Background] Ludwig S, Stier H, Weykam S. Evaluation of Blood Alcohol Concentrations after Oral Administration of a Fixed Combination of Thyme Herb and Primrose Root Fluid Extract to Children with Acute Bronchitis. Drug Res (Stuttg). 2016 Feb;66(2):69-73. doi: 10.1055/s-0034-1398543. Epub 2015 Feb 17. PMID 25823507
- [Background] Kamin W, Maydannik VG, Malek FA, Kieser M. Efficacy and tolerability of EPs 7630 in patients (aged 6-18 years old) with acute bronchitis. Acta Paediatr. 2010 Apr;99(4):537-43. doi: 10.1111/j.1651-2227.2009.01656.x. Epub 2010 Jan 11. PMID 20070280
- [Background] Gruenwald J, Graubaum HJ, Busch R. Evaluation of the non-inferiority of a fixed combination of thyme fluid- and primrose root extract in comparison to a fixed combination of thyme fluid extract and primrose root tincture in patients with acute bronchitis. A single-blind, randomized, bi-centric clinical trial. Arzneimittelforschung. 2006;56(8):574-81. doi: 10.1055/s-0031-1296754. PMID 17009838
- [Background] Kardos P, Bittner CB, Seibel J, Abramov-Sommariva D, Birring SS. Effectiveness and tolerability of the thyme/ivy herbal fluid extract BNO 1200 for the treatment of acute cough: an observational pharmacy-based study. Curr Med Res Opin. 2021 Oct;37(10):1837-1844. doi: 10.1080/03007995.2021.1960493. Epub 2021 Aug 13. PMID 34340607
- [Background] Kemmerich B, Eberhardt R, Stammer H. Efficacy and tolerability of a fluid extract combination of thyme herb and ivy leaves and matched placebo in adults suffering from acute bronchitis with productive cough. A prospective, double-blind, placebo-controlled clinical trial. Arzneimittelforschung. 2006;56(9):652-60. doi: 10.1055/s-0031-1296767. PMID 17063641
- [Background] Haidvogl M, Heger M. Treatment effect and safety of EPs 7630-solution in acute bronchitis in childhood: report of a multicentre observational study. Phytomedicine. 2007;14 Suppl 6:60-4. doi: 10.1016/j.phymed.2006.11.014. Epub 2006 Dec 20. PMID 17184982
- [Background] Matthys H, Kamin W, Funk P, Heger M. Pelargonium sidoides preparation (EPs 7630) in the treatment of acute bronchitis in adults and children. Phytomedicine. 2007;14 Suppl 6:69-73. doi: 10.1016/j.phymed.2006.11.015. Epub 2006 Dec 20. PMID 17184981